CLINICAL TRIAL: NCT06773689
Title: The Role of Cerebral and Peripheral Near-infrared Spectroscopy in Determining Intraoperative Blood Loss in Cancer Surgery
Brief Title: The Role of Near-infrared Spectroscopy Measurements in Determining İntraoperative Blood Loss in Cancer Surgery
Status: Completed | Type: Observational
Sponsor: Dr Abdurrahman Yurtaslan Ankara Oncology Training and Research Hospital (Other)
Responsible Party: Principal Investigator, Ozlem Sen, Doctor, Dr Abdurrahman Yurtaslan Ankara Oncology Training and Research Hospital
Other Study IDs: 2015-01/01
Record Dates: First submitted 2025-01-03; First posted 2025-01-14 (Actual); Last update posted 2025-01-14 (Actual); Status verified 2025-01

CONDITIONS: Near-Infrared Spectroscopy; Cancer Surgery

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Major cancer surgeries often involve significant intraoperative blood loss and require transfusion. Conventional markers, such as hemoglobin (Hb) and hematocrit (Hct), provide limited insight into tissue oxygenation and transfusion thresholds. Near-infrared spectroscopy (NIRS) is a non-invasive approach for monitoring regional tissue oxygen saturation and guiding transfusion decisions. This study aimed to evaluate the role of cerebral (cSO₂) and peripheral (pSO₂) NIRS measurements in identifying intraoperative blood loss and determining transfusion thresholds during major cancer surgeries.

DETAILED DESCRIPTION:
This prospective observational study included 65 patients aged 18-75 years who underwent major cancer surgery. cSO₂ and pSO₂ were monitored at three time points: baseline (T1), pre-transfusion or significant blood loss (T2), and the end of surgery (T3).Hemodynamic parameters, acid-base status, hemoglobin levels, estimated blood loss, and transfusion volumes were recorded.Patients were divided into transfused (group 1) and non-transfused (group 2) cohorts. Statistical analyses included t-tests, Mann-Whitney U tests, and receiver operating characteristic (ROC) analysis.

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anesthesiologists (ASA) physical status I-III
* major cancer surgery in the General Surgery, Urology, and Obstetrics and Gynecology departments

Exclusion Criteria:

* carotid artery stenosis
* recent myocardial infarction
* history of cerebrovascular events
* prior neck surgery,
* cervical disc herniation
* spinal cord injury,
* sudden vision loss,
* deep vein thrombosis,
* refusal to participate.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Sixty-five adult patients (aged 18-75 years) with American Society of Anesthesiologists (ASA) physical status I-III who were scheduled for major cancer surgery in the General Surgery, Urology, and Obstetrics and Gynecology departments
Sampling Method: Non-Probability Sample
Enrollment: 65 (Actual)
Dates: Start 2015-01-01 (Actual); Primary Completion 2015-05-01 (Actual); Study Completion 2015-09-30 (Actual)

PRIMARY OUTCOMES:
cerebral NIRS measurements | T1 (Baseline): Before the start of surgery T2 (Pre-transfusion / Abundant bleeding): In the event of significant blood loss or just before transfusion T3 (At the end of surgery; assessed up to 5 minutes)
  Near-infrared spectroscopy
peripheral NIRS measurements | T1 (Baseline): Before the start of surgery T2 (Pre-transfusion / Abundant bleeding): In the event of significant blood loss or just before transfusion T3 (At the end of surgery; assessed up to 5 minutes)
  Near-infrared spectroscopy

SECONDARY OUTCOMES:
Hemoglobin | T1 (Baseline): Before the start of surgery T2 (Pre-transfusion / Abundant bleeding): In the event of significant blood loss or just before transfusion T3 (At the end of surgery; assessed up to 5 minutes
  İntraoperative blood loss
Hematocrit | T1 (Baseline): Before the start of surgery T2 (Pre-transfusion / Abundant bleeding): In the event of significant blood loss or just before transfusion T3 (At the end of surgery; assessed up to 5 minutes
  intraoperative blood loss
Estimated Blood Loss | T1 (Baseline): Before the start of surgery T2 (Pre-transfusion / Abundant bleeding): In the event of significant blood loss or just before transfusion T3 (At the end of surgery; assessed up to 5 minutes
  intraoperative blood loss